CLINICAL TRIAL: NCT07254702
Title: Prospective Safety Cohort Study VLA1553-406
Brief Title: Prospective Safety Cohort Study After VLA1553 Vaccination in Municipalities Selected for Participation in the VLA1553 Pilot Vaccination Strategy in Brazil
Status: Enrolling by invitation | Type: Observational
Sponsor: Valneva Austria GmbH (Industry)
Collaborators: Fundação Butantan (Unknown); Coalition for Epidemic Preparedness Innovations (Other)
Responsible Party: Sponsor
Other Study IDs: VLA1553-406
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Chikungunya Virus Infection
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Biological: Live-attenuated CHIKV vaccine VLA1553 — Non-interventional study: VLA1553 is used in the pilot vaccination strategy which will start along with this observational study.

SUMMARY:
This is an observational study with primary data collection, which will combine a prospective safety cohort study and an SCRI study.

DETAILED DESCRIPTION:
This prospective safety cohort study will be conducted in selected Brazilian municipalities participating in a pilot vaccination strategy. A total of 5,000 participants will be recruited. The primary objective is to estimate the incidence rates of a predefined set of AEs which constitute safety concerns. The secondary objectives are to measure the relative risk associated with VLA1553 administration for a predefined set of AEs which constitute safety concerns, and to assess the frequency of occurrence of any collected AE which are medically attended or meet the criteria of seriousness This study also aims to investigate VLA1553's safety in underrepresented populations by collecting all AEs, not just AEs which constitute safety concerns.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female participants who received a single dose of VLA1553 at a vaccination unit while participating in the pilot vaccination strategy.
2. Individuals that are target for the pilot vaccination strategy at the time of vaccination.
3. Individuals understanding and being able to comply with all scheduled follow-up calls/contacts and study procedures.
4. Have given informed consent/assent prior to entering the study.

Exclusion Criteria:

1. Individuals who have received investigational products within the 30 days prior to VLA1553 vaccination, or individuals who have received VLA1553/IXCHIQ previously or any authorized or approved CHIKV vaccine.
2. Individuals residing outside of the study municipalities or are not expected to remain in the study municipalities for the next 24 weeks after vaccination.
3. Pregnant women: women exposed to VLA1553 anytime during their pregnancy or within 30 days preceding their last menstrual period will be invited to participate in a separate pregnancy surveillance study (study identifier VLA1553-403).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This study will collect data from approximately 5,000 individuals who received VLA1553, as per label, as part of the pilot vaccination strategy in selected municipalities in Brazil.
Sampling Method: Non-Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2026-02-02 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2027-02-28 (Estimated)

PRIMARY OUTCOMES:
To estimate the incidence rates of a predefined set of AEs which constitute safety concerns according to the VLA1553 Risk Management Plan following the administration of the live-attenuated VLA1553 vaccine | From enrollment until Day 60
  For each safety concern, the risk windows after VLA1553 administration are defined as:
  1. 30 days for Chikungunya-like adverse reactions;
  2. 60 days for cardiac events, choosing a more conservative window than the 42 days suggested by the Brighton Collaboration recommendations on myocarditis;
  3. 60 days for arthritis to account for late-onset or potentially immune-mediated cases

SECONDARY OUTCOMES:
To measure the relative risk associated with VLA1553 administration for a predefined set of AEs which constitute safety concerns as per the VLA1553 Risk Management Plan for those AEs that have a defined risk window following vaccination. | From enrollment until Day 120
To assess the frequency of occurrence of predefined AEs which are medically attended or meet the criteria of seriousness. | From enrollment until Month 6
  1. Frequency of occurrence of predefined chronic chikungunya-like adverse reactions;
  2. frequency of predefined SAEs;
  3. frequency of occurrence of arthralgia;
  4. frequency of occurrence of prolonged arthralgia;
  5. frequency of predefined CHIKV infection symptoms;
  6. frequency of occurrence of predefined chronic CHIKV infection symptoms

OTHER OUTCOMES:
To assess the frequency of occurrence of AEs (not exclusively those of safety concern) following VLA1553 vaccination when co-administered or concomitantly administered with other vaccines. | From enrollment until Month 6
To assess the frequency of occurrence of AEs (not exclusively those of safety concern) in populations underrepresented or excluded in clinical trials with VLA1553. | From enrollment until Month 6
  1. Individuals aged ≥ 65 years old (including those with chronic medical conditions);
  2. individuals with acute or progressive, unstable, or uncontrolled clinical conditions;
  3. individuals with autoimmune or inflammatory disorders (including with impaired or dysregulated immune responses);

CONTACTS AND LOCATIONS:
Locations (4):
- Brazil (4):
  - Universidade Federal Do Ceará, Fortaleza, Ceará
  - Universidade Federal de Minas Gerais, CT Terapias Avançadas e Inovadoras, Belo Horizonte, Minas Gerais
  - Centro de Pesquisas Clínicas Universidade Federal Sergipe, Hospital e Maternidade São João de Deus, Laranjeiras, Sergipe
  - Fundação Faculdade Regional De Medicina De São José Do Rio Preto, São Pedro, São Paulo

IPD SHARING:
Plan to Share IPD: Undecided